CLINICAL TRIAL: NCT05819242
Title: The Reliability And Validity Of A Smartphone App For Measuring Wrist And Metacarpophalangeal Joint Motion
Brief Title: The Reliability And Validity Of A Smartphone App
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ömer Faruk ÖZÇELEP, Researcher, Kirsehir Ahi Evran Universitesi
Other Study IDs: AEUFTR
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis; Carpal Tunnel Syndrome
Keywords: reliability; validity; range of motion
MeSH Terms: conditions — Arthritis, Rheumatoid; Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Adults
  Interventions: Diagnostic Test: Angulus
- Rheumatoid Arthritis
  Interventions: Diagnostic Test: Angulus
- Carpal Tunnel Syndrome
  Interventions: Diagnostic Test: Angulus

INTERVENTIONS:
Diagnostic Test: Angulus — Smartphone app

SUMMARY:
The goal of this observational study is to validate a smartphone app called Angulus. The main question it aims to answer is:

• Is an Angulus App valid and reliable system for masuring hand and wrist range of motion?

Participants will be evaluated by goniometers which is a gold standart for range of motion assessment.

ELIGIBILITY:
Inclusion Criteria:

* a history of previous traumatic hand or wrist injury in the upper extremity,
* pain in the hand and wrist during evaluation
* orthopedic, neurologic, or rheumatologic disease

Exclusion Criteria:

* not to understand the command that the therapist give

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Range of Motions | 15 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code